CLINICAL TRIAL: NCT01544829
Title: The Acute Effect of 2 Different Serving Regimens of Theobromine on Theobromine Concentration in the Blood & Physiological Effects
Brief Title: The Acute Effect of 2 Different Serving Regimens of Theobromine on Physiological Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-SCC-0465
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Cardiovascular Diseases
Keywords: theobromine; heart rate; blood lipids
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Theobromine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Comparator: Single serving of theobromine (Active Comparator)
  Interventions: Dietary Supplement: Theobromine
- Multiple servings of theobromine (Active Comparator)
  Interventions: Dietary Supplement: Theobromine
- Placebo capsules (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Theobromine — Single dose of theobromine
  Arms: Active Comparator: Single serving of theobromine
Dietary Supplement: Theobromine — Multiple doses of theobromine
  Arms: Multiple servings of theobromine
Dietary Supplement: Placebo — Placebo capsules
  Arms: Placebo capsules

SUMMARY:
The main aim of this study is to determine whether there is a difference in the physiological effects of theobromine when provided via a single serving compared to multiple servings adding up to the same amount of theobromine provided on a day.

This study also aims to study the pharmacokinetics of theobromine after administration once per day versus administration 4 times per day.

Hypothesis: the effects on heart rate are less pronounced when a high dose of theobromine is given in 4 smaller doses.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and post-menopausal women: no medical conditions which might affect study measurements (judged by study physician)
* Age 40-70 years
* BMI ≥ 18 and ≤ 30 kg/m2
* Blood pressure, heart rate, haematological and clinical chemical parameters within the normal reference range as judged non clinically significant by research physician
* Written informed consent

Exclusion Criteria:

* Previous cardiovascular event(s) (stroke, TIA, angina, myocardial infarction, heart failure)
* Diabetes mellitus
* Reported weight loss or gain of 10% body weight or more during a period of 6 months prior to screening
* Reported intense sporting activities > 10 h/week
* Use of over-the -counter prescribed medication which may interfere with study measurements, as judged by the physician
* Use of antibiotics in the three months before screening or during the run-in period.
* Currently smoking or being a non-smoker for less than 6 months and reported use of any nicotine containing products in the 6 months preceding the study and during the study itself
* High caffeine consumption: reported consumption of more than 8 cups/cans of caffeine-containing drinks per day, i.e. coffee, black or green tea and cola (also cola light, diet & zero) OR consumption of more than 1 energy drink per day

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Heart rate | 3 days
  Measured during 24h (every 15 minutes during the day and every 30 minutes during the night) for 3 periods

SECONDARY OUTCOMES:
Blood pressure | Measured during 24h (every 15 minutes during the day and every 30 minutes during the night) for 3 periods
Hematocrit | Measured on day 1 and 2 (at time points -5min and 24h) for 3 periods
Serum blood lipids | Measured on day 1 and 2 (at time points -5min and 24h) for 3 periods
Serum glucose and insulin concentrations | Measured on day 1 and 2 (at time points -5min, 3h, 5h, 10h and 24h) for 3 periods

CONTACTS AND LOCATIONS:
Overall Officials: Wieneke Koppenol, MSc, Study Director — Unilever R&D
Locations (1):
- Eurofins Optimed, Gières, France